CLINICAL TRIAL: NCT03857295
Title: Clinical and Microbiological Analyses of Infections Following NeuroSurgery: a Retrospective, Single-center Study
Brief Title: Infections Following NeuroSurgery (INS)
Acronym: INS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Alessandra Oliva, Principal Investigator, Neuromed IRCCS
Other Study IDs: IDAO_1
Record Dates: First submitted 2019-02-22; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Infections Nervous System; Nosocomial Infection; Bacterial Infections; Antibiotic Resistant Infection
Keywords: infections; neurosurgery; multi drug resistance; spondylodiscitis; sepsis
MeSH Terms: conditions — Cross Infection; Bacterial Infections; Infections; Discitis; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventions — No intervention

SUMMARY:
Neurosurgery (NS) is essential for the treatment of various diseases such as malignant tumors, vascular conditions, spinal stenosis or trauma. However, NS can be complicated by the onset of infections, directly related to surgery or to hospitalization.

Little is known regarding the epidemiology, the optimal treatment regimens and the outcome of infections following NS (I-NS).

The study aims at investigating the clinical and microbiological characteristics as well as the outcomes of I-NS occurring at a single Institution (IRCCS Neuromed, Pozzilli, Italy) during the period 2016-2018.

Patients with at least 1 infective episode requiring antimicrobial therapy are included in this retrospective observational study.

DETAILED DESCRIPTION:
Neurosurgery (NS) is essential for the treatment of various diseases such as malignant tumors, vascular conditions, spinal stenosis or trauma. However, one of the major complication is the occurrence of infections following NS (I-NS), with reported rate between 0.5% and 15% depending on the type of NS and the presence/absence of foreign bodies (i.e ventricular shunts, brain stimulators, spinal fixation systems).

I-NS might be related to NS and include meningitis, brain abscesses or spinal infections; I-NS might be also related to the hospitalization and include nosocomial pneumonia, bloodstream and urinary tract infections, especially in elder and frail patients.

While risk factors have been investigated in several studies, little is known about the epidemiology, the optimal treatment regimens and the outcomes of I-NS.

The knowledge of the causative agents of I-NS and the local epidemiology might lead to an early initiation of an appropriate and definite antimicrobial therapy, with obvious consequences in terms of treatment failure and mortality reduction, in line with antimicrobial stewardship principles. Moreover, being aware of the outcomes of I-NS might allow the comprehension of the risk factors associated with clinical cure, recurrence or mortality.

Based on these premises, the principal aim of this single-center, retrospective, observational study is to evaluate the clinical and microbiological characteristics as well as the outcomes of I-NS observed at IRCCS Neuromed (Pozzilli, Italy) over the 2016-2018 period.

Secondary aims are:

i) to analyze the clinical and microbiological characteristics based on the different types of I-NS (i.e. meningitis, brain abscesses, spinal infections, nosocomial pneumonia, bloodstream infections, urinary tract infections); ii) to investigate the presence of multi-drug resistance of the causative agents of I-NS; iii) to correlate the antimicrobial treatment regimens with the observed outcomes of I-NS (i.e. clinical cure, recurrence of infections at 6 months, 30-days mortality).

Patients hospitalized at IRCCS Neuromed with at least 1 infective episode requiring antimicrobial therapy between 2016-2018 will be included in the study. Data will be collected from patient records and will be anonymously registered in an electronic database.

The following data will be collected: type of infection (defined in in accordance with international guidelines); general characteristics of patients (age, gender, type and number of NS, reason for NS, comorbidities); clinical presentation of I-NS (sepsis/septic shock); laboratory and radiological data; microbiological characteristics of I-NS (causative agents; antimicrobial susceptibility profile); antimicrobial therapy (type and number of antimicrobials, length of therapy, empiric versus definite therapy); outcome (30-days mortality, clinical cure, 6-months recurrence of infection)

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized at IRCCS Neuromed between 2016-2018
* Patients with at least 1 infective episode
* Patients receiving antimicrobial therapy

Exclusion Criteria:

* Patients with incomplete data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized at IRCCS Neuromed with at least 1 infective episode requiring antimicrobial therapy between 2016-2018 will be included in the study. Data will be collected from patient records and will be anonimously registered in an electronic database.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-03-11 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with sepsis/septic shock | From the date of inclusion until the date of sepsis/septic shock diagnosis, assessed up to 6 months
  Sepsis or septic shock at the onset of infection Sepsis includes a life-threatening condition and organ dysfunction induced by a disregulated host response to infection (change ≥2 points in SOFA) and septic shock includes persisting hypotension requiring vasopressors to maintain MAP≥65 mmHg AND serum lactate levels ≥2mmol/L despite adequate liquid support.
  Collected measurement data will be aggregated as follows: no sepsis/sepsis/septic shock
Number of participants with multi-drug resistant microorganisms | From the date of inclusion until the date of antimicrobial susceptibility report availability, assessed up to 6 months
  Presence of resistance to >3 class of antimicrobials, as it appears in the antimicrobial susceptibility report.
  Collected measurement data will be aggregated as follows: presence/absence of multi-drug resistance
mortality | 30-days
  Evaluation of mortality of patient with infection.

SECONDARY OUTCOMES:
Correlation of the antimicrobial treatment regimens with the observed outcomes of I-NS | 6-months
  Correlation of the antimicrobial treatment regimens with the observed outcomes of I-NS
Number of participants with Recurrence of infection | 6-months
  Return of the same infection after an infection-free period

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Oliva, MD, PhD, Principal Investigator — IRCCS Neuromed

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Renz N, Ozdirik B, Finger T, Vajkoczy P, Trampuz A. Infections After Cranial Neurosurgery: Prospective Cohort of 103 Episodes Treated According to a Standardized Algorithm. World Neurosurg. 2018 Aug;116:e491-e499. doi: 10.1016/j.wneu.2018.05.017. Epub 2018 May 30. PMID 29758368
- [Background] Riordan MA, Simpson VM, Hall WA. Analysis of Factors Contributing to Infections After Cranioplasty: A Single-Institution Retrospective Chart Review. World Neurosurg. 2016 Mar;87:207-13. doi: 10.1016/j.wneu.2015.11.070. Epub 2015 Dec 22. PMID 26721616
- [Background] Conen A, Fux CA, Vajkoczy P, Trampuz A. Management of infections associated with neurosurgical implanted devices. Expert Rev Anti Infect Ther. 2017 Mar;15(3):241-255. doi: 10.1080/14787210.2017.1267563. Epub 2016 Dec 13. PMID 27910709
- [Background] Chen F, Deng X, Wang Z, Wang L, Wang K, Gao L. Treatment of severe ventriculitis caused by extensively drug-resistant Acinetobacter baumannii by intraventricular lavage and administration of colistin. Infect Drug Resist. 2019 Jan 21;12:241-247. doi: 10.2147/IDR.S186646. eCollection 2019. PMID 30718963
- [Background] McClelland S 3rd, Hall WA. Postoperative central nervous system infection: incidence and associated factors in 2111 neurosurgical procedures. Clin Infect Dis. 2007 Jul 1;45(1):55-9. doi: 10.1086/518580. Epub 2007 May 21. PMID 17554701
- [Background] Lener S, Hartmann S, Barbagallo GMV, Certo F, Thome C, Tschugg A. Management of spinal infection: a review of the literature. Acta Neurochir (Wien). 2018 Mar;160(3):487-496. doi: 10.1007/s00701-018-3467-2. Epub 2018 Jan 22. PMID 29356895
- [Background] Rutges JP, Kempen DH, van Dijk M, Oner FC. Outcome of conservative and surgical treatment of pyogenic spondylodiscitis: a systematic literature review. Eur Spine J. 2016 Apr;25(4):983-99. doi: 10.1007/s00586-015-4318-y. Epub 2015 Nov 19. PMID 26585975
- [Background] Li YD, Wong CB, Tsai TT, Lai PL, Niu CC, Chen LH, Fu TS. Appropriate duration of post-surgical intravenous antibiotic therapy for pyogenic spondylodiscitis. BMC Infect Dis. 2018 Sep 17;18(1):468. doi: 10.1186/s12879-018-3377-1. PMID 30223785
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338